CLINICAL TRIAL: NCT01563770
Title: A Double Blind, Randomized Placebo-controlled Cross-over Study on the Cardiovascular Effects of Salvia Miltiorrhiza Extract (Danshen) in Patients With Hypertension and Hyperlipidemia.
Brief Title: Cardiovascular Effects of Salvia Miltiorrhiza Extract (Danshen)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: QPHT-35
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-01

CONDITIONS: Dyslipidemias; Hypertension; Vasodilation; Oxidative Stress; Inflammation
Keywords: Hyperlipidemia; Hypertension; Vasodilation; Oxidative stress; Inflammation; Hemostasis; Hemorheology; Cardiovascular diseases; Cardiovascular agents; Salvia miltiorrhiza; Danshen; Danshen root extract; Molecular Mechanisms of Pharmacological Action; Therapeutic Uses
MeSH Terms: conditions — Dyslipidemias; Hypertension; Aneurysm; Inflammation; Hyperlipidemias; Cardiovascular Diseases | interventions — dan-shen root extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Salvia miltiorrhiza extract (Danshen) (Experimental): p.o. Salvia miltiorrhiza extract, 1.5 g twice daily for four consecutive weeks
  Interventions: Dietary Supplement: Salvia miltiorrhiza extract
- placebo (Placebo Comparator): p.o. placebo, twice daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Salvia miltiorrhiza extract — 3 capsules of 500 mg Salvia miltiorrhiza extract, twice daily for four consecutive weeks
  Other Names: Danshen
  Arms: Salvia miltiorrhiza extract (Danshen)
Dietary Supplement: Placebo — 3 placebo capsules, twice daily for four consecutive weeks
  Arms: placebo

SUMMARY:
Rationale: Extracts of the plant Salvia miltiorrhiza (Danshen) have been used as traditional Chinese medicine in the treatment of cardiovascular diseases, such as angina pectoris and myocardial infarction. Several preclinical studies point towards promising effects of Danshen on risk factors of atherosclerotic cardiovascular diseases, such as hyperlipidemia and hypertension.

Objective: Our primary objective is to determine the effect of Salvia miltiorrhiza extract (Danshen) on hyperlipidemia. Secondary objective is to investigate the effect of Danshen on hypertension. Further objectives are to determine its effect on endothelial function, oxidative stress, inflammation, hemostasis and hemorheology, and on insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-70
* Women:

  * postmenopausal, or
  * use of contraceptive pill
* Hyperlipidemia:

  * elevated level of triglycerides: > 1.7 mmol/L, or
  * elevated level of LDL-cholesterol: > 3.5 mmol/L
* Hypertension:

  * systolic pressure > 140 mm Hg, or
  * diastolic pressure > 90 mm Hg
* Signed informed consent

Exclusion Criteria:

* Alcohol or drug abuse
* History of cardiovascular disease (myocard infarct, angina pectoris, CVA)
* Diabetes mellitus, when treated with insulin
* Pregnancy
* Hyperlipidemia which needs conventional treatment

  * elevated level of triglycerides: > 8 mmol/L
  * elevated level of LDL-cholesterol: > 5 mmol/L
* Hypertension which needs conventional treatment:

  * systolic pressure > 180 mm Hg
  * diastolic pressure > 110 mm Hg
* Clinically significant liver disease (3 times the upper normal limit of ALAT,ASAT)
* Clinically significant anemia (male Hb < 6,9 mmol/L, female < 6,25 mmol/L)
* Renal disease defined as MDRD < 60 ml/min/1.73m2
* Participation to any drug-investigation during the previous 90 days
* Use of any herbal product during the previous 30 days
* Concomitant (chronic) use of:

Medicinal products:

* ACE-inhibitors, including a.o. captopril, enalapril, ramipril
* AT1-antagonists, including a.o. losartan, valsartan, irbesartan
* Statins, including a.o. simvastatin, rosuvastatin
* Anticoagulant drugs, including a.o. aspirin
* Calciumantagonists (including a.o. amlodipine, nifedipine, verapamil)
* Use of more than 1 antihypertensive drug
* High-dose antihypertensive medication (above defined daily dose)
* Drugs which are exclusively metabolised by CYP3A4 (Flockhart DA; P450 drug interaction table, including a.o. erythromycin, midazolam, cyclosporine, HIV antivirals)

Food products:

* (Antioxidant) vitamin supplements
* Other herbs, including a.o. St John's wort
* Grapefruit juice

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Hyperlipidemia | after 4 weeks of treatment with Danshen
  Blood tests: lipids, in particular LDL-cholesterol.

SECONDARY OUTCOMES:
Hypertension | after 4 weeks of treatment with Danshen
Endothelial function | after 4 weeks of treatment with Danshen
Plasma markers of oxidative stress | after 4 weeks of treatment with Danshen
Vascular inflammation and inflammatory activation of adipose tissue | after 4 weeks of treatment with danshen
Hemostasis and hemorheological parameters | after 4 weeks of treatment with Danshen
Insulin sensitivity | after 4 weeks of treatment with Danshen

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD, PhD, Professor, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] van Poppel PC, Breedveld P, Abbink EJ, Roelofs H, van Heerde W, Smits P, Lin W, Tan AH, Russel FG, Donders R, Tack CJ, Rongen GA. Salvia Miltiorrhiza Root Water-Extract (Danshen) Has No Beneficial Effect on Cardiovascular Risk Factors. A Randomized Double-Blind Cross-Over Trial. PLoS One. 2015 Jul 20;10(7):e0128695. doi: 10.1371/journal.pone.0128695. eCollection 2015. PMID 26192328